CLINICAL TRIAL: NCT05264675
Title: Functional Outcome After Suture or EIP-transfer in EPL-rupture After Distal Radius Fracture
Brief Title: Functional Outcome After EPL-rupture After Distal Radius Fracture
Status: Recruiting | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: VGFOUGSB-964048
Record Dates: First submitted 2022-02-18; First posted 2022-03-03 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Distal Radius Fracture
Keywords: EPL-rupture; Distal radius fracture; Function; ADL
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary suture: primary suture of EPL
  Interventions: Procedure: primary suture
- EIP- transfer: transfer of the EIP to EPL
  Interventions: Procedure: EIP-transfer

INTERVENTIONS:
Procedure: primary suture — Primary suture of the EPL-tendon
  Groups: Primary suture
Procedure: EIP-transfer — transfer of the EIP-tendon to the EPL-tendon
  Groups: EIP- transfer

SUMMARY:
Rupture of the extensor pollicis longus, (EPL) is a common complication after distal radius fractures. A rupture prevents the thumb extension, which in turn has a negative impact on hand function. An EPL-rupture can either be surgically treated by primary suture, which means that the ends of the tendon are sutured. This is however not recommended if the tendon is weakened. In such cases the rupture can be treated by a transfer of, most often, extensor indicis proprius (EIP) to the thumb.

Distal radius fractures are common and a rupture of the EPL-tendon is a known complication thar interferes with hand function and therefore more studies on this patient group are warranted.

The aim of this prospective study is to compare regaining of thumb function after surgery, with the non-injured side, after primary suture and EIP-transfer after EPL-rupture as a complication following distal radius fracture.

DETAILED DESCRIPTION:
Rupture of the long extensor tendon of the thumb (extensor pollicis longus, EPL) is a common complication after distal radius fracture. The incidence has been shown to be about 1% after surgical treatment of the fracture and up to 5% after non-surgical treatment.

The reason why the tendon ruptures after minimally displaced fractures may be reduced blood flow to the tendon. After surgical treatment of a fracture, the cause of rupture may be irritation of the tendon caused by the osteosynthesis material. A rupture means that the thumb cannot be extended, which affects the function of the hand negatively.

EPL rupture can either be operated with primary suture, which means that the ends of the tendon are found and sutured, however this is not recommended if the tendon is weakened, for example due to poor vascularisation. In such a case, the EPL rupture can be repaired by moving a tendon, (usually the extensor indicis proprius, EIP), to the thumb .

Previous studies focusing on function after EPL rupture have been small and have not differentiated EPL ruptures with different underlying causes and the regimen of post-operative care has not been uniform.

Since distal radius fracture is a very common injury and rupture of the EPL tendon is a known complication that affects hand function, it is important that more studies are done on this patient group. Function should be evaluated both with objective and patient-related outcome measures. Knowledge of function after surgery is important for patients, surgeons and rehabilitation staff.

Purpose

The purpose of the present prospective study is to compare recovery of thumb function relative to the non-injured side after primary suture and EIP transfer respectively in rupture of the EPL after distal radius fracture.

Questions

How do patients rate their function after primary suture or EIP transfer?

How much recovery of thumb function occurs relative to the non-injured hand?

Do the groups differ in these respects?

Intervention

After primary suture/tendon transfer and cast immobilization (4 weeks after primary suture and 2 weeks after tendon transfer, respectively), patients will begin exercise according to a specific exercise program for thumb mobility. Between training sessions, an individually adapted, static splint is used with the thumb in extension (2 weeks after primary suture and 4 weeks after tendon transfer, respectively).

Six weeks postoperatively, free mobilization is allowed in light activities of daily living with progressively increased load and training according to the program continues.After twelve weeks, the patient has no restrictions regarding load.

Data collection will take place at 3 and 6 months postoperatively,

The grouping will be based on the treatment method chosen by the surgeon as this is related to the nature of the injury.

Power calculation

A power calculation was made based on the assumption that the group has a mean QuickDASH score of 25 points (SD 8) preoperatively and that the difference between the groups would be 6.8 points, which corresponds to "minimal clinically important difference". To reach a power of 0.80 with alpha 0.05, 22 patients per group are needed. To compensate for a presumed dropout, 30 patients per group are planned to be included.

The patients will be selected via the planning system for operations. The inclusion is expected to last for up to two years.

Data processing

Grip and pinch strength and mobility will be calculated as a percentage of the non-injured side and an average of the percentage will be calculated. Any statistical difference between operated and non-operated side and between the groups will be calculated with t-test.

Expected result / Clinical significance

The expected result is that the patients regain a large part of their function, which is of great importance for the individual patient, no difference between the groups is expected to emerge.

The study is expected to confirm that the treatment regimens used work well, which is important as Sahlgrenska University Hospital strives to use evidence-based treatment methods.

ELIGIBILITY:
Inclusion criteria:

* Distal Radius Fracture
* EPL-rupture

Exclusion Criteria:

* comorbidity interfering with thumb function
* inability to fill in forms

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with distal radius fractures who suffer from rupture of the EPL-tendon
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
range of motion | 3 months postoperatively
  extension, flexion, abduction, retroposition of thumb
range of motion | 6 months postoperatively
  extension, flexion, abduction, retroposition of thumb

SECONDARY OUTCOMES:
strength | 3 months postoperatively
  pinch, lateral pinch, grip strength
strength | 6 months postoperatively
  pinch, lateral pinch, grip strength

OTHER OUTCOMES:
Quick-DASH (Disabilities of the Arm, Shoulder and Hand) | 3 months postoperatively
  Patient rating of function. Minimum score 0 points, maximum score 100 points. Higher scores indicate a worse outcome.
Quick-DASH (Disabilities of the Arm, Shoulder and Hand) | 6 months postoperatively
  Patient rating of function. Minimum score 0 points, maximum score 100 points. Higher scores indicate a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Andreasson, Md Dr, Principal Investigator — Sahlgrenska Universitetssjukhuset
Locations (1):
- Sahlgrenska University Hospital, Mölndal, Sweden

IPD SHARING:
Plan to Share IPD: No